CLINICAL TRIAL: NCT01026987
Title: A Pilot Study of G-CSF +/- Plerixafor (AMD3100) Mobilized Donor CD34+ Enriched Peripheral Blood Mononuclear Cells for the Treatment of Allogeneic Stem Cell Transplant Recipients With Limited Donor Engraftment
Brief Title: Granulocyte Colony-stimulating Factor (G-CSF) Plus or Minus AMD3100 for Engraftment Post Allogeneic Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-1824 / 201011859
Record Dates: First submitted 2009-12-01; First posted 2009-12-07 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Stem Cell Transplant Patients
MeSH Terms: interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; plerixafor; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Related Donors: G-CSF & AMD3100 (Experimental): G-CSF 10 ug/kg SC daily for 5 days. AMD3100 320 mcg/kg IV over 30 min on Day 5. Leukapheresis on Day 5.
  Interventions: Drug: G-CSF; Drug: AMD3100; Procedure: Leukapheresis
- Recipient (Other): Stem Cell Infusion on Day 0
  Interventions: Procedure: Stem Cell Infusion

INTERVENTIONS:
Drug: G-CSF — Unrelated donors will receive only G-CSF (10 ug/Kg S/C qDay x5-6 days) prior to pheresis (collection of the stem cells). Unrelated donors will only be followed per NMDP guidelines.
  Other Names: Neupogen
  Arms: Related Donors: G-CSF & AMD3100
Drug: AMD3100
  Other Names: Plerixafor; Mozobil
  Arms: Related Donors: G-CSF & AMD3100
Procedure: Leukapheresis
  Arms: Related Donors: G-CSF & AMD3100
Procedure: Stem Cell Infusion
  Arms: Recipient

SUMMARY:
Patients who have not had adequate blood count recovery post related or unrelated stem cell transplant will be given a "boost" of T-cell depleted, enriched stem cells to hopefully improve their blood counts.

DETAILED DESCRIPTION:
Patients who have not had adequate blood count recovery post related or unrelated stem cell transplant will be given a "boost" of T-cell depleted, enriched stem cells to hopefully improve their blood counts.

The unrelated donors will receive G-CSF prior to pheresis (collection of the stem cells) to boost the number of CD34+ cells. The related donors will receive G-CSF and AMD3100 prior to pheresis to boost the number of CD34+ cells. Once the CD34+ cells are collected they will be T-cell depleted using a cell separation device called the CliniMACS systems. The CliniMACS system will select the CD34+ cell and remove the T-cells. By removing the T-cells we can minimize the risk of Graft Versus Host Disease (GVHD). The enriched CD34+ cells will be given to them to hopefully give them a "boost" of cells that can permanently produce new blood cells to improve their risk of infection and bleeding.

ELIGIBILITY:
Inclusion Criteria:

Recipient

* Must be age ≥ 18
* Must have ≥90 % donor cells in the unfractionated peripheral blood based on either XY FISH or standard STR.
* More than 60 days post allogeneic stem cell transplantation.
* Must meet one of the following criteria:
* platelets < 20,000 or
* ANC<500 or
* transfusion dependent for at least one cell line and /or
* on growth factor support (G-CSF) without adequate response for 30 days and
* no reversible etiology found after an allogeneic stem cell transplantation
* Patient has an ECOG performance status of 0-2.
* The original stem cell donor must be available, willing, and medically able to undergo Mobilization and a maximum of 2 apheresis procedures
* Each patient (recipient) or legal guardian and donor must be willing to participate as a research subject and must sign an informed consent form.

Unrelated Donors

* NMDP guidelines for eligibility will be followed using G-CSF alone mobilization.

Related donors

* Must be ≥18 yrs old and ≤ 75 years old.
* Donor must be sero-negative for HIV-1&2 antibody and HTLV-I&II antibody, by FDA licensed test.
* Donor must have adequate renal function as defined by serum creatinine ≤ 1.5X institution ULN and AST and ALT ≤ 3X ULN and total bilirubin less than 2 mg/dl.
* Donor must be agreeable to mobilization and the second donation of PBMC.
* Women of child bearing potential should be willing to avoid becoming pregnant while receiving treatment with plerixafor.
* Donor must have adequate peripheral venous catheter access for leukapheresis or must agree to placement of a central catheter.

Exclusion Criteria:

Recipient

* Patients with confirmed relapse of their original disease
* Participation in other clinical trials that involve investigational drugs or devices except with permission from the Principal Investigator and Sponsor.
* Patients with documented active viral, bacterial or fungal infections.
* Documented allergy to murine proteins or iron dextran.
* Pregnancy
* Patients with immune mediated graft dysfunction.

Donor

* Evidence of active infection at the time of study entry.
* Medical or physical reason which makes the donor unlikely to tolerate or cooperate with growth factor therapy and leukapheresis
* Factors which place the donor at increased risk for complications from leukapheresis or G-CSF therapy(e.g., autoimmune disease, multiple sclerosis, sickle cell trait, coronary artery disease).
* Pregnancy (positive serum or urine beta-HCG) or breastfeeding. Women of childbearing age must avoid becoming pregnant while on the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-04-29 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2016-06-08 (Actual)

PRIMARY OUTCOMES:
Time to neutrophil engraftment | 100 days post CD34+ selected, T-Cell depleted transplant
  For recipients with ANC < 500 or growth factor support dependent at study entry, Time to neutrophil improvement is measured from the date of CD34+ selected, T-Cell depleted infusion to the first of 3 consecutive measurements of neutrophil count > 500/μl without growth factor support for >7 days prior.
  RBC transfusion engraftment - independence from RBCs without growth factors.
Time to platelet engraftment | 100 days post CD34+ selected, T-Cell depleted transplant
  For recipients with platelets < 20,000 or platelet transfusion dependent at study entry, Time to platelet improvement is measured from the date of CD34+ selected, T-Cell depleted infusion to the of 3 consecutive measurements of platelet count ≥ 20,000/ul without platelet transfusion support for 7 days.
Time to red blood cell (RBC) improvement | 100 days post CD34+ selected, T-Cell depleted transplant
  For recipients who are RBC transfusion dependent at study entry, Time to RBC improvement is measured from the date of CD34+ selected, T-Cell depleted infusion to the first date of hemoglobin >9.0g/dL without > 1 RBC transfusion during the previous 56 days.

SECONDARY OUTCOMES:
To assess the feasibility of collecting adequate donor CD34+ enriched T-cell depleted peripheral blood stem cells using G-CSF+ plerixafor from related donors and G-CSF alone from unrelated donors. | Day 0 (transplant day)
Toxicities associated with the CD34+ collection (donors) | 30 days post mobilization
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Phenotypically and functionally characterize donor CD34+ and donor T-cells mobilized by G-CSF from unrelated donors and mobilized with G-CSF + plerixafor from related donors. | Day of mobilization (Day 0)
Overall survival (recipients) | 1 year from date of transplant
  Overall survival is the time from the date of CD34+ selected, T-Cell depleted infusion to death.
Incidence and severity of acute Graft vs Host Disease (GVHD) | 100 days post-transplant
  Incidence and severity of acute GVHD will be assessed based on the Seattle criteria
Toxicities associated with CD34+ cell infusion (recipients) | 30 days post-transplant
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Disease-free survival | 1 year from date of transplant
  Disease-Free survival is the time from the date of CD34+ selected, T-Cell depleted infusion to disease relapse or death.
Incidence and severity of acute Graft vs Host Disease (GVHD) | 2 years post-transplant
  Incidence and severity of chronic GVHD will be assessed based on the Seattle criteria
Rate of transplant-related mortality (TRM) | 100 days post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: John DiPersio, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu